CLINICAL TRIAL: NCT00748150
Title: A Phase II, Open-Label, Uncontrolled, Single Center Study to Evaluate Safety and Immunogenicity of Flu Vaccine Influenza Vaccine (Surface Antigen, Inactivated) Ph.Eur, Formulation 2008-2009, When Administered to Non-Elderly Adult and Elderly Subjects
Brief Title: Safety and Immunogenicity of Influenza Vaccine (Surface Antigen, Inactivated) Ph.Eur, Formulation 2008-2009, When Administered to Non-Elderly Adult and Elderly Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V78P6S; 2008-000939-17
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Influenza
Keywords: flu; influenza; influenza vaccine antigen; immunogenicity; antibody response; intra muscular; elderly; non-elderly
MeSH Terms: conditions — Influenza, Human | interventions — Antigens, Surface

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Flu Vaccine Influenza Vaccine (Surface Antigen, Inactivated) Ph.Eur, Formulation 2008-2009

INTERVENTIONS:
Biological: Flu Vaccine Influenza Vaccine (Surface Antigen, Inactivated) Ph.Eur, Formulation 2008-2009 — 1 dose, 0.5 mL of Flu Vaccine Influenza Vaccine (Surface Antigen, Inactivated) Ph.Eur, Formulation 2008-2009

SUMMARY:
Annual trial for registration influenza vaccine with the strain composition for season 2008/2009

DETAILED DESCRIPTION:
At enrolment, subjects were stratified into two age strata (18 to 60 years, over 60 years). Total duration of the study is three weeks. Vaccinations were to be administered on day 1. Blood samples were collected at day 1 (baseline, before the vaccination) and at day 22 (three weeks after the vaccination). Sera were tested by Hemagglutination Inhibition (HI) assay. Safety was assessed until 3 weeks after the vaccination.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age, mentally competent, willing and able to give informed consent prior to study entry
* available for all the visits scheduled in the study and able to comply with all study requirements
* in good health as determined by:

  1. medical history
  2. physical examination
  3. clinical judgment of the investigator

Exclusion Criteria:

* Any serious (in the judgment of the investigator) disease including, but not limited to:

  1. Cancer, except for localized skin cancer
  2. Advanced congestive heart failure
  3. Chronic obstructive pulmonary disease (COPD
  4. Autoimmune disease (including rheumatoid arthritis)
  5. Acute or progressive hepatic disease
  6. Acute or progressive renal disease
  7. Severe neurological or psychiatric disorder
  8. Severe asthma
* History of any anaphylactic reaction and/or serious allergic reaction following a vaccination, a proven hypersensitivity to any component of the study vaccine (e.g. to ovalbumin, chicken protein, chicken feathers, influenza viral protein, neomycin, polymixin)
* Known or suspected (or have a high risk of developing) impairment/alteration of immune function (excluding that normally associated with advanced age) resulting for example from:

  1. Receipt of immunosuppressive therapy (any parenteral or oral corticosteroid or cancer chemotherapy/radiotherapy) within the past 60 days and for the full length of the study
  2. Receipt of immunostimulants,
  3. Receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within the past 3 months and for the full length of the study,
  4. Suspected or known HIV infection or HIV-related disease.
* Known or suspected history of drug or alcohol abuse.
* The subject has a bleeding diathesis or condition associated with prolonged bleeding time that in the investigator's opinion would interfere with the safety of the subject
* Women who are pregnant or woman of child-bearing potential unwilling to practice acceptable contraception for the duration of the study (21 days).
* Influenza vaccination or laboratory confirmed influenza within the last 6 months and more than one influenza vaccination within the past 12 months
* Within the past 4 weeks, the subject has received:

  1. another vaccine
  2. any investigational agent
* Any acute or chronic infection requiring systemic antibiotic treatment or antiviral therapy within the last 7 days.
* The subject has experienced an acute exacerbation of a COPD within the past 14 days
* The subject has experienced fever (i.e. axillary temperature ³ 38.0°C) within the last 3 days
* Severely obese with Body Mass Index (BMI) > 35 kg/m2
* Any condition, which, in the opinion of the investigator, might prevent the subject from participation or interfere with the evaluation of the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of antibody response to each influenza vaccine antigen, as measured by haemagglutination inhibition (HI) test on Day 0 and on Day 21 | 21 days

SECONDARY OUTCOMES:
Evaluation of safety of the influenza vaccine | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- The Health Centre, Heath Road, Woolpit, Bury Saint Edmunds, Suffolk, United Kingdom